CLINICAL TRIAL: NCT06372873
Title: Deep Learning-enabled Ultrasound Classification of Anterior Talofibular Ligament Injury in China: A Retrospective, Multicentre, Diagnostic Study
Brief Title: Deep-learning For Ultrasound Classification of Anterior Talofibular Ligament Injury
Status: Active, not recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Zhu Jiaan, Chairman, Peking University People's Hospital
Other Study IDs: 2023PHB211-001
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Deep Learning; Ultrasound; Anterior Talofibular Ligament

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group I: mild-strain injury of ATFL
  Interventions: Other: re-evaluate by two senior radiologists in our medical center
- Group II: partial ligament tears of ATFL
  Interventions: Other: re-evaluate by two senior radiologists in our medical center
- Group III: complete rupture of ATFL
  Interventions: Other: re-evaluate by two senior radiologists in our medical center
- Group IV: avulsed fractures
  Interventions: Other: re-evaluate by two senior radiologists in our medical center

INTERVENTIONS:
Other: re-evaluate by two senior radiologists in our medical center — The allocated images obtained from the contributing hospitals will be re-evaluated by two senior radiologists in our clinical center

SUMMARY:
Ultrasound (US) is a more cost-effective, accessible, and available imaging technique to assess anterior talofibular ligament (ATFL) injuries compared with magnetic resonance imaging (MRI). However, challenges in using this technique and increasing demand on qualified musculoskeletal (MSK) radiologists delay the diagnosis. Using datasets from multiple clinical centers, the investigators aimed to develop and validate a deep convolutional network (DCNN) model that automates classification of ATFL injuries using US images with the goal of providing interpretable assistance to radiologists and facilitating a more accurate diagnosis of ATFL injuries.

The investigators collected US images of ATFL injuries which had arthroscopic surgery results as reference standard form 13 hospitals across China;Then the investigators divided the images into training dataset, internal validation dataset, and external validation dataset in a ratio of 8:1:1; the investigators chose an optimal DCNN model to test its diagnostic performance of the model, including the diagnostic accuracy, sensitivity, specificity, F1 score. At last, the investigators compared the diagnostic performance of the model with 12 radiologists at different levels of expertise.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old
* patients who had experienced an first-episode, acute ankle sprain and received US examination within 14 days post injury
* patients who had a corresponding arthroscopic surgery result for classification of the ATFL injury.

Exclusion Criteria:

* patients who had a previous history of ankle open trauma or ankle joint surgery
* there were any soft-tissue or bone tumors in the ankle
* there was concurrent with any other rheumatoid arthritis
* the image quality was low or there were severe artifacts (eg, anisotropic artifacts)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: As mentioned above
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate whether the US images are in consensus with the ATFL injury classification of the reference standard | Baseline
  The radiologists in our clinical center will re-evaluate whether the US images are in consensus with the classification of ATFL injury of its reference standard

CONTACTS AND LOCATIONS:
Overall Officials: Jiaan Zhu, Dr, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gribble PA, Bleakley CM, Caulfield BM, Docherty CL, Fourchet F, Fong DT, Hertel J, Hiller CE, Kaminski TW, McKeon PO, Refshauge KM, Verhagen EA, Vicenzino BT, Wikstrom EA, Delahunt E. Evidence review for the 2016 International Ankle Consortium consensus statement on the prevalence, impact and long-term consequences of lateral ankle sprains. Br J Sports Med. 2016 Dec;50(24):1496-1505. doi: 10.1136/bjsports-2016-096189. Epub 2016 Jun 3. PMID 27259753
- [Background] Colo G, Bignotti B, Costa G, Signori A, Tagliafico AS. Ultrasound or MRI in the Evaluation of Anterior Talofibular Ligament (ATFL) Injuries: Systematic Review and Meta-Analysis. Diagnostics (Basel). 2023 Jul 10;13(14):2324. doi: 10.3390/diagnostics13142324. PMID 37510068
- [Background] Cao M, Liu S, Zhang X, Ren M, Xiao Z, Chen J, Chen X. Imaging diagnosis for anterior talofibular ligament injury: a systemic review with meta-analysis. Acta Radiol. 2023 Feb;64(2):612-624. doi: 10.1177/02841851221080556. Epub 2022 Mar 27. PMID 35343253
- [Background] Gao Y, Zeng S, Xu X, Li H, Yao S, Song K, Li X, Chen L, Tang J, Xing H, Yu Z, Zhang Q, Zeng S, Yi C, Xie H, Xiong X, Cai G, Wang Z, Wu Y, Chi J, Jiao X, Qin Y, Mao X, Chen Y, Jin X, Mo Q, Chen P, Huang Y, Shi Y, Wang J, Zhou Y, Ding S, Zhu S, Liu X, Dong X, Cheng L, Zhu L, Cheng H, Cha L, Hao Y, Jin C, Zhang L, Zhou P, Sun M, Xu Q, Chen K, Gao Z, Zhang X, Ma Y, Liu Y, Xiao L, Xu L, Peng L, Hao Z, Yang M, Wang Y, Ou H, Jia Y, Tian L, Zhang W, Jin P, Tian X, Huang L, Wang Z, Liu J, Fang T, Yan D, Cao H, Ma J, Li X, Zheng X, Lou H, Song C, Li R, Wang S, Li W, Zheng X, Chen J, Li G, Chen R, Xu C, Yu R, Wang J, Xu S, Kong B, Xie X, Ma D, Gao Q. Deep learning-enabled pelvic ultrasound images for accurate diagnosis of ovarian cancer in China: a retrospective, multicentre, diagnostic study. Lancet Digit Health. 2022 Mar;4(3):e179-e187. doi: 10.1016/S2589-7500(21)00278-8. PMID 35216752